CLINICAL TRIAL: NCT06217172
Title: Use of the Multidimensional Health Assessment Questionnaire (MDHAQ/RAPID3) in Follow-up of Patients With Rheumatoid Arthritis by Telemedicine: A Non-Inferiority Randomized Clinical Trial
Brief Title: RHEUPP - A Rheumatological Follow-up Management App
Acronym: RHEUPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: PANLAR - 2023 Innovation Award (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2023-0057
Record Dates: First submitted 2023-12-29; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; telehealth; mhealth app
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultrasonography; High-Energy Shock Waves; ametantrone

STUDY DESIGN:
Intervention Model Description: Number of participants was considered after sample size estimation for non-inferiority margins to the outcome expected.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Other): RHEUPP App follow-up
  Interventions: Device: RHEUPP App
- Control Group (Other): Usual follow-up
  Interventions: Other: Usual Follow-up

INTERVENTIONS:
Device: RHEUPP App — RHEUPP App; Monthly RAPID3 response; General recommendations for managing Flare through App and Social Monitor for appropriate orientation; 3 month consultation by telehealth.
  Other Names: Other analysis: X-Ray (Sharp van der Heijde Score); Ultrasound (US10 Score); Laboratory tests; SF-36; SUS; ASES-8; eHEALS; HAQ; FACIT; FIQ; FSQ; HAQ; MDHAQ
  Arms: Intervention Group
Other: Usual Follow-up — Usual Care in Rheumatoid Arthritis Ambulatory Service
  Other Names: Other analysis: X-Ray (Sharp van der Heijde Score); Ultrasound (US10 Score); Laboratory tests; SF-36; SUS; ASES-8; eHEALS; HAQ; FACIT; FIQ; FSQ; HAQ; MDHAQ
  Arms: Control Group

SUMMARY:
The purpose of this Non-inferiority Randomized Clinical Trial is to evaluate the effectiveness of RHEUPP App during telehealth follow-up in a population of Rheumatoid Arthritis patients from a Tertiary Rheumatology Service in South Brazil.

The main question[s] it aims to answer are:

• Using RHEUPP App in telemedicine is not inferior to usual care in terms of means obtained by CDAI.

Participants will be stratified by CDAI and then randomized 1:1 for intervention or control group. They will be evaluated at study starting, in 3 and 6 months, an extended evaluation after 12 months of recruitment is predicted.

Researchers will compare intervention and control group to detect differences between usual care and Telehealth follow-up and determine if the last is not less effective in our study population of rheumatic patients.

DETAILED DESCRIPTION:
Participants with access to digital media will be sent a weblink for accessing the study's electronic questionnaires by electronic message or email, with a maximum interval of one week before or after your in-person consultation, according to the research participant's preference. A tablet will be made available to patients who choose to carry out the survey on the day of their in-person assessment. Participants randomized to the intervention group will receive guidance regarding the download or access to the RHEUPP application, with a period of training and adaptation to the tool, to be carried out by Social Monitor.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18y or older)
* Rheumatoid Arthritis according to the 2010 EULAR/ACR criteria
* Access to digital media (electronic messages, e-mail)

Exclusion Criteria:

* Other rheumatological diseases (except Sjögren's Syndrome)
* Inability to understand the instrument in general or assistance from third parties (family member or caregiver) in carrying out the questionnaire at a disadvantage
* Incomplete information in data collection
* Patients with changes in their treatment in the last 4 weeks or treatment change plan at recruitment to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of telehealth monitoring according to differences in means of CDAI | From study start to 26 weeks (extended evaluation at 52 weeks)
  Non-inferiority margin of -0.6 u.m defined based on a 50% of Good EULAR Response criteria (with a 10% increase for possible losses and refusals, this number should be 88). The calculation considered a non-inferiority margin of -6 u.m., a power of 80%, level of significance of 5%, difference of 0 u.m between the means and standard deviation of 10.6 u.m. (data
  Non-inferiority margin of -6 u.m defined based on a 50% of Good EULAR Response criteria

SECONDARY OUTCOMES:
Non-inferiority of telehealth monitoring according to differences in means of DAS28 | From study start to 26 weeks (extended evaluation at 52 weeks)
  Non-inferiority margin of -0.6 u.m defined based on a 50% of Good EULAR Response criteria
Differences in means of SDAI between groups | From study start to 26 weeks (extended evaluation at 52 weeks)
  Simplified Disease Activity Index for Rheumatoid Arthritis (SDAI) is calculated as follows: [SDAI = SJC + TJC +PGA + EGA + CRP]. Remission is defined as an SDAI of <3.3, low disease activity as ≤11, moderate disease activity as ≤26 and high disease activity as >26.
Response rate to ACR20 | From study start to 26 weeks (extended evaluation at 52 weeks)
  The ACR20 is a composite measure defined as an improvement of 20% in the number of tender and swollen joints and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Response rate to ACR50 | From study start to 26 weeks (extended evaluation at 52 weeks)
  The ACR50 is a composite measure defined as an improvement of 50% in the number of tender and swollen joints and a 50% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Response rate to ACR70 | From study start to 26 weeks (extended evaluation at 52 weeks)
  The ACR70 is a composite measure defined as an improvement of 70% in the number of tender and swollen joints and a 70% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP).
Changes in baseline for DAS28 | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  The Disease Activity Score-28 for Rheumatoid Arthritis (DAS28) range from 0 to 9.4 and are calculated using tender joints, swollen joints, general health, and a laboratory measure of acute inflammation.
Changes in baseline for CDAI | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  The Clinical Disease Activity Index (CDAI) is based on the simple summation of the count of swollen/tender joint count of 28 joints along with patient and physician global assessment on VAS (0-10 cm) Scale for estimating disease activity. The CDAI has range from 0 to 76
Changes in baseline for SDAI | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  The Simplified Disease Activity Index for Rheumatoid Arthritis (SDAI) is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), patient and physician global assessment of disease activity [visual analogue scale (VAS) 0-10 cm] and level of C-reactive protein (mg/dl, normal <1 mg/dl). The SDAI has a range from 0 to 100.
Percentage of participants achieving remission criteria by DAS28, CDAI and SDAI | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Based on the definition of remission criteria by ACR/EULAR for each score
Percentage of participants achieving remission criteria by ACR/EULAR | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Based on the definition of remission criteria by ACR/EULAR for each score
Percentage of participants dropping-out from study | From study start to 26 weeks (extended evaluation at 52 weeks)
  Estimation based on absolute number of participants
Change from baseline in Physician and Patient Global Assessment (PGA-VAS) | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  PGA is often assessed by a single question with a 0-10 or 0-100 response. The content can vary and relates either to global health (e.g., how is health overall) or to disease activity (e.g., how active is arthritis).
Change from baseline in RAPID3 and its correlations | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  RAPID3 is a composite index of physical function, pain and PGA-VAS each scored 0-10, comprising a 0-30 score. Higher scores indicate poorer status. Four RAPID3 severity categories have been proposed: high (>12), moderate (6.1-12), low (3.1-6) and near remission (≤3).
Change from baseline in MDHAQ and its correlations | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Multi-dimensional health assessment questionnaire (MDHAQ) - PMID 16273781 [Authorized License from RWS Life Sciences]
Change from baseline to System Usability Scale (SUS) and its correlations | From study start to 26 weeks (extended evaluation at 52 weeks)
  System Usability Scale (SUS): Lewis JR, Sauro J. The factor structure of the system usability scale. In: Lecture Notes in Computer Science (including subseries Lecture Notes in Artificial Intelligence and Lecture Notes in Bioinformatics) 94-103; 2009.
Change from baseline to uMARS and its correlations | From study start to 26 weeks (extended evaluation at 52 weeks)
  Based on the Brazilian version DOI: https://doi.org/10.33448/rsd-v12i6.42056
Change from baseline to ASES-8 Questionnaire and its correlations | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Measure by the Brazilian version of ASES-8 https://doi.org/10.1590/1516-3180.2018.0354071218
Change from baseline to HAQ and its correlations | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Health Assessment Questionnaire (HAQ) is a tool for measuring functional status in rheumatology. Scores of 0 to 1 are generally considered to represent mild to moderate difficulty, 1 to 2 moderate to severe disability, and 2 to 3 severe to very severe disability.
Percentage of participants in the EULAR response criteria for "Good response" and "Moderate Response" | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Based on the definition criteria by ACR/EULAR
Percentage of participants achieving Boolean remission in the ACR/EULAR criteria | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Based on the definition of Boolean remission criteria by ACR/EULAR
Change from baseline in detection of Flare by RAPID3 | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Flare will be considered when the RAPID3 score increases by more than 2 points in relation to the previous score or if the current RAPID3 is greater than 4.
Correlations with clinical assessment and other scores with Flare detection by the score RAPID3 | From study start to 26 weeks (extended evaluation at 52 weeks)
  Flare on RAPID3 score will be considered if increases by more than 2 points in relation to the previous score or if the current RAPID3 is greater than 4.
Assessment of FACIT and its correlations | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  PMID: 15868614
Assessment of FIQ and FSQ scores and its correlations | From study start, 13 weeks and 26 weeks (extended evaluation at 52 weeks)
  Based on the Brazilian version PMID: 23604595 / https://doi.org/10.1186/s42358-020-00139-3
Cost-effectiveness evaluation | From study start to 26 weeks (extended evaluation at 52 weeks)
  To evaluate cost-effectiveness and added value of the instrument in routine assistance, the number of consultations or attendance needs in emergency care/emergency care for participants throughout their follow-up at the study; travel cost estimate; evaluation of the score result in the decision professional's therapy and user's perception of the use of the instrument in monitoring your rheumatological disease.

CONTACTS AND LOCATIONS:
Overall Officials: Claiton V Brenol, Prof.PhD, Principal Investigator — Federal University of Health Science of Porto Alegre

REFERENCES:
- [Background] Lineburger IB, Brenol CV, Goularte AS, Pinheiro EP, Hirakata VN. Cross-cultural and clinical validation of the MDHAQ/RAPID3 questionnaire in electronic format for a Brazilian population of patients with rheumatoid arthritis. Adv Rheumatol. 2022 Nov 22;62(1):46. doi: 10.1186/s42358-022-00278-9. PMID 36419141
- See also: Citation of PANLAR Award Recipient for the project development. — https://www.panlar.org/en/articulo/winners-2023-panlar-awards